CLINICAL TRIAL: NCT06321354
Title: Pre-emptive Infiltration of the Scalp with Diprospan Plus Ropivacaine for Pain After Craniotomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-066-02-3
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pain; Postoperative Children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The diprospan plus ropivacaine group (Experimental): Patients in the diprospan plus ropivacaine group will receive a peri-incisional scalp infiltration with 15ml diprospan and 15mg of 1% ropivacaine and normal saline miscible liquids.
  Interventions: Drug: The diprospan plus ropivacaine group
- The ropivacaine group (Active Comparator): Patients in the ropivacaine group will receive a peri-incisional scalp infiltration with 15mg of 1%
  Interventions: Drug: The ropivacaine group

INTERVENTIONS:
Drug: The diprospan plus ropivacaine group — The local infiltration solution containing 0.5ml diprospan and 15mg of 1% ropivacaine. The total volume is 30 ml. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Arms: The diprospan plus ropivacaine group
Drug: The ropivacaine group — The local infiltration solution containing 15mg of 1% ropivacaine. The total volume is 30 ml. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Arms: The ropivacaine group

SUMMARY:
At present, pediatric postoperative analgesia has not been fully understood and controlled, particularly craniotomy surgery. On the one hand, professional evaluation of postoperative pain for young children is difficult; on the other hand, the particularity of craniotomy adds (such as consciousness obstacle, sleepiness, et al) disturbance to the pain assessment in children. Although opioids administration is regarded as the first-line analgesic for post-craniotomy pain management, it may be associated with delayed awakening, respiratory depression, hypercarbia and it may interfere with the neurologic examination. For the avoidance of side-effects of systemic opioids, local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was unsatisfactory due to its short pain relief duration, steroid as adjuvant can enhance postoperative analgesia and prolong postoperative analgesia time. As is reported that postoperative pain of craniotomy is mainly caused by skin incision and reflection of muscles, preventing the liberation of inflammatory mediators around the incision seems to be more effective than simply blocking nerve conduction. Researchers have clarified that the addition of diprospan to local infiltration of analgesia could provide significant analgesic effects and significantly prolong the duration of analgesic effects without obvious complications for various types of surgeries. To date, no studies have evaluated the addition of diprospan to local infiltration for patients receiving craniotomy.

Thus, investigators suppose that pre-emptive scalp infiltration with steroid (Diprospan) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in children.

ELIGIBILITY:
Inclusion Criteria:

* An elective craniotomy under general anesthesia; American Society of Anesthesiologists (ASA) physical status of I or II; Participates with an anticipated fully recovery within 2 hours postoperatively; Informed consent by parent(s) and/or legal guardian.

Exclusion Criteria:

* History of allergies to any of the study drugs; Drugs with confirmed or suspected sedative or analgesic effects; receiving any painkiller within 24 h before surgery; children who received steroids; Psychiatric disorders; Uncontrolled epilepsy; Chronic headache; Peri-incisional infection; Body mass index exceeded the 99th percentile for age; Children who must use a patient-controlled analgesia (PCA) device; Children who cannot understand an instruction of pain scales before surgery

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
modified Children's Hospital of Eastern Ontario Pain Scale (mCHEOPS) | At 24 hours after the operation
  Postoperative pain will be estimated by using the modified Children's Hospital of Eastern Ontario Pain Scale (mCHEOPS). 0 indicates no pain, 10 indicates the most severe pain imaginable.

SECONDARY OUTCOMES:
modified Children's Hospital of Eastern Ontario Pain Scale (mCHEOPS) | At 2 hours, 4 hours, 8 hours, 48 hours, 72 hours, 1 week after surgery
  Postoperative pain will be estimated by using the modified Children's Hospital of Eastern Ontario Pain Scale (mCHEOPS). 0 indicates no pain, 10 indicates the most severe pain imaginable.
The time to the first rescue analgesic | Within 48 hours after the operation
  Rescue analgesics will be administered if the patient exhibits signs of sympathetic stimulation in the form of undue tachycardia, a rise in mean arterial pressure (rise of >20% from the baseline), and mCHEOPS score above 5 (range 1 to 10) or if the children are in obvious pain and distress at any time point during a subjective assessment by the intensivist or parents.
Patient satisfactory scale (PSS) | At 2 hours, 4 hours, 8 hours, 48 hours, 72 hours, 1 week after surgery
  0 for unsatisfactory, and 10 for very satisfied
Length of stay (LOS) | Approximately 1 weeks after the operation
  LOS will be recorded as the number of nights spent in hospital after surgery.
The occurrence of postoperative nausea and vomiting (PONV) | At 2 hours, 4 hours, 8 hours, 24 hours after surgery
  PONV will be rated by participants as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay Sedation Scale (RSS) | At 2 hours, 4 hours, 8 hours, 24 hours after surgery
  1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
The occurrence of respiratory depression | Within 48 hours after the operation
  Respiratory depression is defined as persistent (more than 1 minutes) oxygen desaturation 90 percent or respiratory rate less than 8 breaths per minute, or oxygen desaturation less than 94 percent along with respiratory rate less than 10 breaths per minute requiring supplemental oxygen to maintain oxygen saturation more than 94 percent in the absence of clinically obvious upper airway obstruction.
Heart rate | During the operation and at 2 hours, 4 hours, 8 hours, 24 hours after surgery
Mean arterial pressure | During the operation and at 2 hours, 4 hours, 8 hours, 24 hours after surgery
The total consumption of opioids during the operation | During procedure
The total consumption of anaesthetic during the operation | During procedure
Wound Healing Score | At 1 month after surgery
  Skin Healing 1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection 1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth 1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable
Incisional related adverse events | Approximately 1 weeks after the operation
  Incisional related adverse events Including delayed incisional healing, incisional infection, intracranial infection, scar healing.
The occurrence of the Adverse events (AEs) and serious adverse events (SAEs) | Within 1 weeks after the operation
  An AE was defined as any untoward medical occurrence. An SAE included death, immediately life-threatening conditions, coma, in-patient hospitalisation or prolongation of existing hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Fang, M.D, Principal Investigator — Beijing Tiantan Hospital; Ge Ming, M.D, Principal Investigator — Beijing Children's hospital affiliated to capital medical university
Locations (2):
- China (2):
  - Beijing Children's hospital affiliated to capital medical university, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.